CLINICAL TRIAL: NCT04448249
Title: Advanced Practice Nurse Intervention Versus Usual Care for Hypertension Control: Study Protocol for an Open-label Randomized Controlled Trial
Brief Title: Advanced Practice Nurse Intervention Versus Usual Care for Hypertension Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hotel Dieu University Hospital, France (Other)
Responsible Party: Principal Investigator, Jacques Blacher, MD, PhD, Hotel Dieu University Hospital, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APN
Record Dates: First submitted 2020-06-16; First posted 2020-06-25 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
Keywords: Advanced Pratice Nurse; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The interventional group keeps a traditional follow up (day hospitalization then consultation with a MD within two to twelve months) but also meets an APN between the day hospitalization and the MD consultation, within one to six months
  Interventions: Behavioral: APN intervention
- Control group (No Intervention): The control group of patients keeps a traditional follow-up: day hospitalization then consultation with a MD within two to twelve months

INTERVENTIONS:
Behavioral: APN intervention — APN intervention is divided into five main steps:
  * clinical and paraclinical examinations,
  * appraisal of patient's knowledge,
  * health education on hypertension and treatments,
  * setting a written medication plan with the patient to invest him in his management with adjusting or renewing treatments identically if necessary,
  * decision-making balance between the benefits and risks of non-adherence to medication. A time is scheduled at the end of the intervention to let the patient ask questions or express his difficulties if he needs to.
  Arms: Interventional group

SUMMARY:
Hypertension is the most frequent chronic pathology in France and in the world. It is one of the main modifiable cardiovascular risk factors. In France, 50% of treated hypertensives are uncontrolled and only 30% of treated patients are fully adherent to their antihypertensive treatment. Poor adherence to drug treatments is considered as one of the main causes of non-control of hypertension. Since 2018, a new profession has entered the French healthcare system: Advanced Practice Nurses (APN). They have many broad skills, at the interface of nursing and medical exercises. The purpose of this interventional study is to assess the impact of APN on blood pressure (BP) control in the context of usual care of hypertension thanks to a better adhesion of patients and a better therapeutic alliance. The hypothesis formulated is that an individual APN intervention, included in a usual hypertension management, improves BP control.

DETAILED DESCRIPTION:
This study will be a prospective, open-label, randomized 1-to-1 and monocentric trial, conducted at the Diagnosis and Therapeutic Center of the Hôtel-Dieu University Hospital, Assistance Publique - Hôpitaux de Paris, France.

The patients will be recruited during their visit at the day hospitalization of the Diagnosis and Therapeutic Center of Hôtel-Dieu University Hospital, for hypertension-related complications and cardiovascular risk assessment as part of their hypertension management.

Randomization/allocation will be conducted at the last moment before scheduling appointments.

The "usual care" group will keep a traditional follow-up: day hospitalization then consultation with a MD within approximately 2 to 12 months.

The "intervention" group will meet the APN between the day hospitalization and the MD consultation, within 1 to 6 months (Figure 1).

All data will be collected on site, none remotely. All information required by the protocol will be recorded on a case report form. An explanation will be provided for each missing data. The data will be collected as it is obtained and clearly transcribed into the case report form.

The primary outcome measure will be analyzed using a chi-square test. A p value <0.05 will be considered significant. Participants with missing data for this primary outcome will be considered lost to follow-up. For secondary outcome measures, a chi-square test will be used for qualitative variables compared between the two groups. A paired t-tests will be used for the differences of rate of controlled blood pressure between day hospitalization and MD consultation in each group. Non-adherent participants (APN intervention missed for the interventional group) will be considered in the statistical analysis and the rate of non-adherent participants will be mentioned in the results.Correlations between the realization and the quality of home BP monitoring in MD consultation and controlled BP will also be analyzed. No interim analyses are scheduled.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age,
* treated or untreated hypertension,
* can to provide a written informed consent.

Exclusion Criteria:

* age under 18 years old,
* inability to give a free informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of controlled blood pressure in MD consultation (office blood pressure < 140/90 mmHg) | 12 months
  According to the European and International guidelines, the protocol for office BP measurement will be: 5 minutes rest, 3 measurements at one-minute intervals in supine position followed by 3 standing measurements at one-minute intervals for orthostatic hypotension test. Unattended office blood pressure measurement will be conducted thanks to a supervisor (usually a nurse) who will explain the protocol to the patient before letting him rest in a quiet room and thanks to an automatic sphygmomanometer that can print the statement of measures at the end of the monitoring. Blood pressure level will be estimated by the average of the 2 last blood pressure measures in supine position. We will consider that blood pressure is controlled if systolic blood pressure < 140 mmHg and diastolic blood pressure < 90 mmHg.

SECONDARY OUTCOMES:
Rate of home blood pressure monitoring brought to MD consultation | 12 months
  According to the 2020 International Society of Hypertension (ISH) Global Hypertension Practice Guidelines, the protocol for home BP monitoring will be: 3-day monitoring with a cycle of 3 measures every morning and every evening at one-minute intervals, in a sitting position, after 5 minutes of rest and before meals.
Quality of the home blood pressure monitoring brought to MD consultation | 12 months
  The quality will be assessed by the number of measurements (18 measurements over 3 days according to the protocol).
Rate of therapeutic adjustments during the APN intervention | 6 months
  Rate of therapeutic adjustments among the interventional group during the APN intervention.
Indication(s) of therapeutic adjustments during the APN intervention | 6 months
  Rate of therapeutic adjustments due to lack of efficacy and/or intolerance among the interventional group during the APN intervention.
Difference in rates of controlled blood pressure (office blood pressure < 140/90 mmHg) between day hospitalization and MD consultation in each group. | 12 months
  Evolution of the rate of controlled blood pressure between day hospitalization and MD consultation in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette VAY-DEMOUY, Principal Investigator — Hôpital Universitaire Hôtel-Dieu; AP-HP; Université de Paris, France
Locations (1):
- Hôpital Hôtel-Dieu, Paris, France